CLINICAL TRIAL: NCT03096275
Title: Comparison of the Efficacy of Mycophenolate Mofetil Combined With Methotrexate and Cyclophosphamide for the Treatment of Takayasu's Arteritis
Brief Title: Comparison of Mycophenolate Mofetil and Cyclophosphamide for Active Takayasu's Arteritis
Acronym: CommittedTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese SLE Treatment And Research Group (Other)
Collaborators: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Xinping Tian, Professor of Medicine, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCHCSTAR-006
Record Dates: First submitted 2017-03-13; First posted 2017-03-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2021-04

CONDITIONS: Takayasu Arteritis
Keywords: Mycophenolate mofetil; Methotrexate; cyclophosphamide
MeSH Terms: conditions — Takayasu Arteritis | interventions — Glucocorticoids

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to two treatment arms and were treated for 12 months.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MMF+MTX+Glucocorticoids (Experimental): Patients were treated with Glucocorticoids combined with mycphenolate mofetil(MMF) as well as methotrexate(MTX) treatment for 52 weeks and were followed for 52 weeks.
  Interventions: Drug: MMF; Drug: Glucocorticoids; Drug: MTX
- CYC/AZA+Glucocoticoids (Active Comparator): Patients were treated with Glucocorticoids combined with cyclophosphamide(CYC)/azathioprine(AZA) for 52 weeks and were followed for 52 weeks
  Interventions: Drug: CYC; Drug: Glucocorticoids; Drug: AZA

INTERVENTIONS:
Drug: MMF — Patients were treated with Glucocorticoids combined with methotrexate and mycophenolate mofetil
  Other Names: Guangwei
  Arms: MMF+MTX+Glucocorticoids
Drug: CYC — Patients were treated with Glucocorticoids and cyclophosphamide sequentially with azathioprine
  Other Names: huanlinxianan
  Arms: CYC/AZA+Glucocoticoids
Drug: Glucocorticoids — Patients in the experimental group and comparator group were treated with Glucocorticoids and then gradually tapered
  Other Names: qiangdisong
Drug: MTX — Patients in the experimental group are treated with Glucocorticoids combined with MTX and MMF
  Other Names: jiaandieling
  Arms: MMF+MTX+Glucocorticoids
Drug: AZA — Patients in the active comparator group were treated with Glucocorticoids combined with CYC followed by AZA
  Other Names: liuzuopiaoling
  Arms: CYC/AZA+Glucocoticoids

SUMMARY:
Takayasu's arteritis(TAK) is a rare systemic vasculitis which can cause ischemia or inflammation of the involved organs and increase the overall mortality rate.The traditional treatment of TAK is primarily empirical. The most commonly used drugs for treating active TAK are glucocorticosteroids(GC) and immunosuppressants. However, the genital toxicity of CYC has limited its long term use. In a pilot study carried out by the principal investigator of this study has shown that mycophenolate mofetil(MMF) combined with MTX is effective and with few adverse effects. The purpose of this prospective open-label study is to compare the efficacy and safety of GC+MMF+MTX with GC+CYC followed by GC+AZA for the treatment of active TAK. 150 patients with active TAK will be recruited and randomized in a 2:1 ratio to GC+MMF+MTX group and C+CYC and AZA group. Patients were followed for 52 weeks for efficacy and safety assessment.

DETAILED DESCRIPTION:
Takayasu's arteritis(TAK) is a rare systemic vasculitis which mainly involves aorta and its major branches. However,it is more prevalent in countries and areas along the silk road.Young women at child-bearing age is the most prevalent population.It can cause ischemia or inflammation of the involved organs and increase the overall mortality rate.Although it may be lethal in some patients,it is not well studied due to the rareness of the disease.The traditional treatment of TAK is primarily empirical. The most commonly used drugs for treating active TAK are glucocorticosteroids(GC) and immunosuppressants including cyclophosphamide(CYC), methotrexate(MTX) and azathioprine(AZA) etc. However,no of these drugs have been well studied. In addition, the genital toxicity of CYC, the first line medication for active TAK, has become the major limitation for its long term use for a chronic disease like TAK. Therefore, new immunosuppressants with less toxicity,especially with much less genital toxicity and low malignancy risk is essentially necessary. In a pilot study carried out by the principal investigator of this study has shown that mycophenolate mofetil(MMF) combined with MTX is effective and with few adverse effects. The purpose of this prospective open-label study is to compare the efficacy and safety of GC+MMF+MTX with GC+CYC followed by GC+AZA for the treatment of active TAK. 150 patients with active TAK will be recruited and randomized in a 2:1 ratio to GC+MMF+MTX group and C+CYC and AZA group. Patients were followed for 52 weeks to assess the efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years-old either sex
2. Patients with signed informed consent
3. Fulfill the 1990 ACR Classification Criteria for TAK
4. Patients with active disease according to GACTA criteria

Exclusion Criteria:

1. Prior adverse events when treated with MTX that resulted in dose reduction or discontinuation;
2. Prior treatment with MMF but failed response to MMF;
3. Prior treatment with CYC but failed response to CYC;
4. Renal dysfunction, defined as the estimated GFR <80% or serum creatinine level higher than 1.5 times of upper normal limit;
5. Severe liver function damage defined by serum ALT or AST higher than 2 times of the upper normal limits;
6. Uncontrolled diabetes melitus;
7. Uncontrolled heart failure at baseline;
8. Active infection including tuberculosis , hepatitis B virus, hepatitis C virus, HIV or bacterial or fungal infection;
9. Active upper GI bleeding in the past 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete remission | 52 weeks
  The proportion of patients who reached the pre-defined criteria of complete remission in both groups

SECONDARY OUTCOMES:
Proportion of patients with partial remission | 52 weeks
  Proportion of patients who reached the pre-defined partial remission criteria of the disease
Safety profile of MMF combined with MTX | 52 weeks
  Proportion of adverse events in both treatment groups
Rate of complications | 52 weeks
  Proportion of patients with complications in both treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Xinping Tian, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (7):
- China (7):
  - Hebei Provincial Hospital, Shijiazhuang, Hebei
  - the Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - Xijing Hospital, Xian, Shanxi
  - Beijing Chaoyang Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Xuanwu Hospital, Beijing
  - General Hospital of Tianjing Medical University, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arend WP, Michel BA, Bloch DA, Hunder GG, Calabrese LH, Edworthy SM, Fauci AS, Leavitt RY, Lie JT, Lightfoot RW Jr, et al. The American College of Rheumatology 1990 criteria for the classification of Takayasu arteritis. Arthritis Rheum. 1990 Aug;33(8):1129-34. doi: 10.1002/art.1780330811. PMID 1975175
- [Result] Goel R, Danda D, Mathew J, Edwin N. Mycophenolate mofetil in Takayasu's arteritis. Clin Rheumatol. 2010 Mar;29(3):329-32. doi: 10.1007/s10067-009-1333-6. PMID 20054700
- [Result] Shinjo SK, Pereira RM, Tizziani VA, Radu AS, Levy-Neto M. Mycophenolate mofetil reduces disease activity and steroid dosage in Takayasu arteritis. Clin Rheumatol. 2007 Nov;26(11):1871-5. doi: 10.1007/s10067-007-0596-z. Epub 2007 Feb 28. PMID 17332971
- [Result] Daina E, Schieppati A, Remuzzi G. Mycophenolate mofetil for the treatment of Takayasu arteritis: report of three cases. Ann Intern Med. 1999 Mar 2;130(5):422-6. doi: 10.7326/0003-4819-130-5-199903020-00013. PMID 10068416
- [Result] Ong LM, Hooi LS, Lim TO, Goh BL, Ahmad G, Ghazalli R, Teo SM, Wong HS, Tan SY, Shaariah W, Tan CC, Morad Z. Randomized controlled trial of pulse intravenous cyclophosphamide versus mycophenolate mofetil in the induction therapy of proliferative lupus nephritis. Nephrology (Carlton). 2005 Oct;10(5):504-10. doi: 10.1111/j.1440-1797.2005.00444.x. PMID 16221103
- [Result] Li J, Yang Y, Zhao J, Li M, Tian X, Zeng X. The efficacy of Mycophenolate mofetil for the treatment of Chinese Takayasu's arteritis. Sci Rep. 2016 Dec 7;6:38687. doi: 10.1038/srep38687. PMID 27924855